CLINICAL TRIAL: NCT05242120
Title: Impact of COVID 19 Pandemic on Anesthesia Resident's Training Program in Cairo University Hospitals. A Cross-sectional Study.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Dina Mahmoud Mohamed, Principal investigator, lecturer of anesthesia and ICU and pain management, Kasr El Aini Hospital
Other Study IDs: MS-531-2021
Record Dates: First submitted 2022-02-15; First posted 2022-02-16 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: COVID-19; Anesthesia
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Residents who completed their residency (class 2013,2014 , 2016, 2017): Residents who completed their residency (class 2013,2014 , 2016, 2017)
  Interventions: Other: Survey to access the impact of COVID 19 on anesthesia residency

INTERVENTIONS:
Other: Survey to access the impact of COVID 19 on anesthesia residency — This is a cross-sectional study using an online survey will be conducted on 75 anesthesia residents in Cairo University hospitals. Invitations were sent to residents' groups on WhatsApp. Study objectives were clearly explained at the beginning of the survey, and the participants were encouraged to roll out the survey to as many physicians as possible. This survey contains 62-question, divided into four main sections

SUMMARY:
In December 2019, a cluster of pneumonia cases, caused by a newly identified βcoronavirus, occurred in Wuhan, China.1 The World Health Organization (WHO) officially named the disease as coronavirus disease 2019 (COVID-19), and the International Committee on Taxonomy of Viruses named the virus as severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2).2 On 11 March 2020, the WHO declared the epidemic of COVID-19 as a pandemic.3 The pandemic crisis prioritises critical care for those coronavirus (COVID-19) patients who have been most profoundly affected, and hospitals, staffing, and working practices have been radically adjusted to accommodate this.4,5 The healthcare industry, in particular, has been overwhelmed by the effect of COVID-19 on healthcare resources. This has been underscored by providers concerned about emotional strain and physical exhaustion, access to personal protective equipment (PPE) and medical equipment, workplace exposure to COVID-19 and disease transmission to family members.6 Physicians are essential for any health-care system and at the frontline defense against the COVID-19 pandemic. They play a crucial role in diagnosis, treatment, prevention of disease spread, and public education during this pandemic. Moreover, they are frequently exposed to infected individuals with COVID-19, making them at higher risk of infection than others.7 Anesthesia is one such specialty whose residents are uniquely at risk of exposure to infection in the operating room or ICU. Residents reported that their learning schedule is distorted in our hospital regarding skills because of increase ICU rotations, cancelled elective surgeries, missing one or two of the major rotations. Also, lecturers were stopped and replaced by E-learning after a long period. Examination schedule was changed and so the research schedule. Infection of the trainees (or a member of a family) had a great emotional and physical impact on them.

COVID-19 will not go away any time soon, and therefore the new balance between service provision and training needs to be agreed in a sensitive way to avoid further frustration amongst trainees. Adaptations to these circumstances have delivered new forms of teaching and supervision.

We design this cross-sectional study and implement a survey that included a 58-question to accomplish the specific aims of the present study through comparisons of two groups of residents and to provide plans for the training programme to be less affected by pandemics.

ELIGIBILITY:
Inclusion Criteria:

* Residents of either sex, in the last year or completed their residency (class 2016, and 2017) in Cairo University hospitals spending 2 years in the pandemic. Residents who completed their residency before the pandemic (class2013, 2014).

Exclusion Criteria:

* Residents who did not pass the first part of residency or who did not complete their residency for any other cause rather than the pandemic.

Ages: 25 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 75 anesthesia residents will be enrolled in this study and will be divided into two groups. Group (A) residents who completed their residency before the pandemic (class 2013, 2014) and group (B) residents that main part of their residency at least 2 years in the pandemic (class 2016, 2017)
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2022-02-20 (Estimated); Primary Completion 2022-05-10 (Estimated); Study Completion 2022-05-30 (Estimated)

PRIMARY OUTCOMES:
To measure the degree of affection of the skills acquired by the residents through the pandemic. | 30 minutes
  This is a cross-sectional study using an online survey will be conducted on 75 anesthesia residents in Cairo University hospitals. Invitations were sent to residents' groups on WhatsApp. Study objectives were clearly explained at the beginning of the survey, and the participants were encouraged to roll out the survey to as many physicians as possible. This survey contains 62-question, divided into four main sections

IPD SHARING:
Plan to Share IPD: Undecided